CLINICAL TRIAL: NCT00257647
Title: Use of SV40 siRNA Vectors to Treat CML
Brief Title: Use of SV40 Vectors to Treat Chronic Myeloid Leukemia (CML)
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Ariella Oppenheim, Hadassah Medical Organization
Other Study IDs: 497169-HMO-CTIL; US Army
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2007-04

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: SV40 vectors carrying siRNA — in vitro only use of gene therapy

SUMMARY:
Chronic myeloid leukemia is a serious disease which is characterized by progression from relatively quiescent stages of the disease to an aggressive phase. Although now there is highly successful medical therapy known as Gleevec (Imatinib), the treatment is not always successful and patients do develop resistance. Those patients have limited treatment options. We are developing a gene therapy model of treatment for this disease using pseudoviral particles to insert molecules of genetic material which would not allow the harmful genes causing the leukemia to function.

DETAILED DESCRIPTION:
A novel methodology that facilitates specific silencing of genes has recently been developed. The method is based on the property of small molecules of nucleic acids (RNA) to specifically repress expression of targeted genes. These small interfering RNA (siRNA) molecules were recently demonstrated to repress, in tissue culture cells, one of the two types of the common fusion genes present in CML patients. Those studies showed that treatment with synthetic siRNA inhibited cell growth and increased the sensitivity to imatinib. These findings offer hope that a novel form of gene therapy based on this strategy may improve the treatment outcome of CML patients, particularly when used in combination with other approaches such as the tyrosine kinase inhibitor imatinib that was mentioned above.

Our group has developed an innovative vector that is most suitable to deliver siRNA molecules into human hematopoietic cells with sufficient efficacy. The vector is based on a monkey virus called simian virus 40 (SV40). The viral coat, or capsid, is produced biosynthetically. It was engineered to self-assemble in the test tube around the nucleic acids of choice, and to deliver this DNA or RNA into target cells. This vector is safer than other available viral vectors since all the viral genetic material is excluded from the final product. The vector does not elicit immune response, thus allowing repeated administration.We will start the project by testing the recently published siRNA molecules against one of the fusion genes, and several alternative siRNA molecules that we will design against the other fusion genes. The molecules will be tested for efficacy in tissue culture cell-lines, by measuring repression of the respective fusion gene, reduction in the level of the tyrosine kinase and inhibition of cell growth. The most effective siRNA molecules will be selected for further studies. The vectors will be tested on cell-lines for gene silencing and cell death as before. At the final stage we will test the best vectors for their efficacy in white blood cells obtained from CML patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CML

Exclusion Criteria:

* Under 18 years old
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CML patients which were seen at Hadassah hospital.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2005-09; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah G Rund, MD, Study Chair — Hadassah Medical Organization; Ariella Oppenheim, PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Rund D, Dagan M, Dalyot-Herman N, Kimchi-Sarfaty C, Schoenlein PV, Gottesman MM, Oppenheim A. Efficient transduction of human hematopoietic cells with the human multidrug resistance gene 1 via SV40 pseudovirions. Hum Gene Ther. 1998 Mar 20;9(5):649-57. doi: 10.1089/hum.1998.9.5-649. PMID 9551613
- [Background] Kimchi-Sarfaty C, Ben-Nun-Shaul O, Rund D, Oppenheim A, Gottesman MM. In vitro-packaged SV40 pseudovirions as highly efficient vectors for gene transfer. Hum Gene Ther. 2002 Jan 20;13(2):299-310. doi: 10.1089/10430340252769815. PMID 11812285